CLINICAL TRIAL: NCT02874911
Title: Coordination Training With Complete Body Video Games in Children and Adults With Degenerative Ataxias
Acronym: Move'n Fun
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Move'n Fun
Record Dates: First submitted 2016-08-12; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Spinocerebellar Ataxia
Keywords: Exergaming; Neurodegenerative diseases; Rare disease; Motor exercises; Training; Spinocerebellar ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias; Neurodegenerative Diseases; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- General training (Experimental): Advanced spinocerebellar disease receive 12 weeks of coordinative training based on commercially available videogames (Product names: Nintendo Wii ®, Microsoft XBOX Kinect®).
  Interventions: Other: General training

INTERVENTIONS:
Other: General training — Advanced spinocerebellar disease receive 12 weeks of coordinative training based on commercially available videogames (Product names: Nintendo Wii ®, Microsoft XBOX Kinect®).

SUMMARY:
Exergame training might offer a novel treatment approach even in largely nonambulatory subjects with multisystemic degenerative spinocerebellar ataxia.

DETAILED DESCRIPTION:
Effective treatments for patients with degenerative spinocerebellar ataxia are scarce. It has recently been shown that intensive coordinative training based on either physiotherapy or exergames (= whole-body controlled videogames; might improve degenerative ataxia, but its effectiveness is still disputed. This situation is even more complicated for degenerative ataxia subjects in advanced disease stages and with high multisystemic disease load. Here, underlying neurodegeneration has progressed to many irreversible states and includes many additional extra-cerebellar systems, making functional plasticity and therapeutic success much less likely. Moreover, intervention outcome assessment in subjects unable to walk freely is more delicate. Correspondingly, nonambulatory ataxia subjects in advanced disease stages are currently often excluded from treatment trials, thus leaving them without prospects of access to novel treatments.

The investigators here hypothesized that exergame training might offer a novel treatment approach even in largely nonambulatory subjects with multisystemic degenerative spinocerebellar ataxia. Using a rater-blinded, intraindividual control study design, the investigators show that an individualized exergame training strategy, tailored to individuals' disease stage, improves postural control and ataxia-specific control functions even in advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Advanced spinocerebellar disease
* Advanced impairments in gait and stance, defined as Scale for Assessment and Rating of Ataxia (SARA) subscore gait ≥3 and stance ≥3, but still able to sit without support >10 seconds, as defined by SARA subscore sitting <3
* Age between 5 and 30 years

Exclusion Criteria:

* Any signs of inflammatory, vascular, malformation, or tumor cerebrospinal (CNS) disease
* Visual loss, hearing disturbances, mental retardation and predominant non-ataxia movement disorders (e.g. predominant spasticity, chorea, parkinsonism)

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Gait | Week 13
  Item 1 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8
Stance | Week 13
  Item 2 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8
Sitting | Week 13
  Item 3 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8
Speech disturbance | Week 13
  Item 4 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8
Finger chase | Week 13
  Item 5 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8
Nose-finger Test | Week 13
  Item 6 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8
Fast alternating hand movements | Week 13
  Item 7 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8
Heel-shin slide | Week 13
  Item 8 of the Scale for the Assessment and Rating of Ataxia (SARA) score; total score made up of item 1 - 8

SECONDARY OUTCOMES:
Goal attainment Score | Week 13
  To capture translation of training effects into subjects' daily living and personally relevant activities
Quantitative movement analysis | Week 13
  Postural stability by quantitative movement analysis, using a motion capture system (Product name: VICON MX).

CONTACTS AND LOCATIONS:
Overall Officials: Synofzik Matthis, PD Dr., Principal Investigator — University Hospital Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schatton C, Synofzik M, Fleszar Z, Giese MA, Schols L, Ilg W. Individualized exergame training improves postural control in advanced degenerative spinocerebellar ataxia: A rater-blinded, intra-individually controlled trial. Parkinsonism Relat Disord. 2017 Jun;39:80-84. doi: 10.1016/j.parkreldis.2017.03.016. Epub 2017 Mar 28. PMID 28365204